CLINICAL TRIAL: NCT02122679
Title: A Randomized Trial Investigating the Effect of Tranexamic Acid on Platelet Aggregation Following Infant Cardiopulmonary Bypass
Brief Title: Tranexamic Acid Effect on Platelet Aggregation Following Infant Cardiopulmonary Bypass
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael Wolf, Assistant Professor of Pediatrics, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00073642
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Heart Defect, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): Receive tranexamic acid in operating room.
  Interventions: Drug: Tranexamic Acid
- Placebo group (Placebo Comparator): Receive placebo in the operating room
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Study group
Drug: placebo
  Arms: Placebo group

SUMMARY:
Tranexamic acid is a relatively safe medicine that is used to help the body develop clots and slow down bleeding after large surgeries. While it has already been shown to work well in adults and older children, there is no information on whether it works, and how it works in children younger than 6 months old. The goal of our study is to try and understand whether and how tranexamic acid works in children younger than 6 months old who are having open heart surgery.

We plan to study tranexamic acid by testing its effect when compared with a placebo. The investigators will use a method called randomization - which means patients who agree to be in the study will be entered into a computer. The computer will randomly assign them to either receive the medicine or the placebo. We will then compare effects on the 2 groups of patients. Our goal is to have 50 patients in each group, or 100 patients total. We will not know whether patients receive tranexamic acid or placebo until we review the data collected at the end of the study.

Tranexamic acid is usually given to patients in the operating room during open heart surgery. During open heart surgery patients require cardio-pulmonary bypass which is a machine that replaces the function of the heart and lungs for a short period of time. This allows surgeons to do surgery on the heart itself without having to worry about it moving during the operation. The bypass machine has lots of tubes to carry the blood around it. When blood comes into contact with the tubing it has a tendency to clot. To prevent this patients are given a blood thinner called heparin. Although heparin prevents clotting in the bypass machine, it can also increase the risk of bleeding when the surgery is over. To reduce this risk patients are given another medicine at the completion of surgery called protamine to try and reverse the effect of the blood thinner, heparin.

Even so bleeding remains a significant problem, especially for babies after open heart surgery. Being on the bypass machine and having a lot of suture (stitches) lines increase that risk. In addition, the bypass machine affects the function of platelets, the main component of the body's clotting system. We often have to replenish blood products after surgery to try and stop the bleeding. Some centers, including we , have used the medicine tranexamic acid to try and help with bleeding after surgery. There have been other studies that show it helps with fibrinolysis, which is another important part of the body's clotting system. However, that part of the clotting system is not well developed in infants and therefore likely does not play an important role in preventing bleeding in that age group.

As such, it may be that tranexamic acid impacts platelet function as well, and it is that effect that helps decrease post-operative bleeding in infants younger than 6 months. This has not been previously studied. In order to study the effect that tranexamic acid has on platelets the investigators are proposing the investigators' research trial. The investigators plan to randomize patients to either receive tranexamic acid or placebo in the operating room as described above. The investigators will then draw a small amount of blood from each patient (total of approximately 1 tablespoon) and send it to a special lab for testing of platelet function. The lab test will help us understand whether the platelets function better when patients receive tranexamic acid instead of placebo.

The investigators will also be monitoring other outcomes related to platelet function. These will include how much bleeding patients have after surgery when they are in the intensive care unit, and how much blood products they require to treat that bleeding. The investigators will also monitor labs that are checked routinely in all patients after open heart surgery. The investigators will also track how long it takes each patient to get off the ventilator and how long they spend in the ICU after surgery. All of this data will help us understand whether tranexamic acid makes a positive impact on outcomes after open heart surgery in infants less than 6 months old.

The current standard of care is quite variable within our institution as well as at other institutions. Some anesthesiologists use tranexamic acid while others elect not to. There is no definitive guideline to its current use. The dosing differs from center to center, and there are some centers that do not use it at all.

The investigators' hope is that the results of this study will help us understand the role tranexamic acid plays in preserving the function of platelets after open heart surgery in young infants, and whether that impact translates into improved outcomes for those patients. Based on the results of our research we hope to develop definitive guidelines for the use of tranexamic acid in the population of infants <6 months old undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Infants ≤ 6 months of age undergoing congenital cardiac surgery with cardiopulmonary bypass
2. Cyanotic and non-cyanotic congenital heart disease are eligible for enrollment
3. No patient will be excluded because of race or ethnicity
4. Parental or legal guardian consent will be obtained for all patients prior to enrollment

Exclusion Criteria:

1. Documented or suspected bleeding or coagulation disorder
2. Documented history of occlusive deep venous or arterial thrombosis
3. Cardiac surgery without cardiopulmonary bypass (i.e. Blalock-Taussig shunt, coarctation of the aorta)
4. The need for mechanical circulatory support within 12 hours following cardiopulmonary bypass including extracorporeal membrane oxygenation.
5. Placement of a ventricular assist device
6. Prior enrollment in this study (Stage II Norwood who had been enrolled at their Stage I operation)
7. Parent or legal guardian unable or unwilling to consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Platelet Aggregation | 1 year
  Measure the effect of tranexamic acid on whole blood platelet aggregation as measured by collagen induced platelet aggregometry.

SECONDARY OUTCOMES:
Postoperative bleeding | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States